CLINICAL TRIAL: NCT01807637
Title: Using Transcranial Direct Current Stimulation to Jump Start Gait Training in Chronic Stroke Patients
Brief Title: Transcranial Direct Current Stimulation for Improving Gait Training in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: University of Central Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 138159; 138159 (Other: University of Arkansas for Medical Sciences)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Stroke; Cerebral Vascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transcranial direct current stim (Experimental): tDCS will be applied using a Soterix constant current stimulator with 5 x 5 cm (25cm2) carbon rubber electrodes (Covidien 664 REFX 2x2) applied to the scalp with 10-20 conductive paste. The anodal electrode will be placed over the lower extremity representation of primary motor cortex of the lesioned hemisphere [established during TMS motor threshold testing (Baseline Testing) and the functional MRI assessment]. The cathodal electrode will be placed over the contralateral motor cortex.
  Interventions: Device: transcranial direct current stim (tDCS)
- sham tDCS (Placebo Comparator): Sham stimulation will be performed by turning the stimulator off after the initial sensory experience (30 seconds).
  Interventions: Device: transcranial direct current stim (tDCS)

INTERVENTIONS:
Device: transcranial direct current stim (tDCS) — During anodal tDCS, participants will receive 20 min at 2mA over motor cortex (with 30 seconds of ramp-up and ramp-down). During sham stimulation the stimulator is turned off.

SUMMARY:
The purpose of this study is to determine if transcranial direct current stimulation (tDCS)applied over the lower extremity motor cortex in conjunction with assisted gait training is effective for improving gait in patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors > 3 months from most recent unilateral, stroke based on clinically or experimentally obtained MRI brain scans and behavioral evidence of stroke (e.g., risk factors, hemiplegia, unilateral sensory impairment, or localized higher cortical dysfunction) by report or in the medical record.
* Age: >21 years of age.
* Complete NIH Stroke Scale.
* Sufficient endurance, motor ability and balance to ambulate at least 10 meters continuously with moderate or less assistance.
* Demonstrate gait impairment during ambulation such that gait instability or inefficient gait patterns [gait pattern manifesting "dragging" or "catching" of the affected toes during swing phase of gait, or use of compensatory strategies such as circumducting the affected limb, vaulting with the unaffected limb or hiking the affected hip to clear the toes] are exhibited.
* Pass the Transcranial Magnetic Stimulation (TMS) Adult Safety Screen (TASS) except for items related specifically to stroke and the treatment for stroke.

Exclusion Criteria:

* Edema, skin breakdown, absent sensation of the affected lower limb which interferes with the peroneal nerve stimulator.
* History of potentially fatal cardiac arrhythmias, such as ventricular tachycardia, supraventricular tachycardia, and rapid ventricular response atrial fibrillation with hemodynamic instability.
* Demand pacemakers or any other implanted electronic systems.
* Pregnant women, uncontrolled seizure disorder, Parkinson's Disease, Spinal cord injury, Traumatic brain injury with evidence of motor weakness, Multiple sclerosis.
* Documented episode in the medical record of a seizure occurring 1 month or more post stroke for which the patient received consultation or treatment for said seizures. Seizures occurring within the first month following a stroke are not exclusionary unless followed by another seizure.
* Fixed ankle plantar flexor contracture, peroneal nerve injury at the fibular head as the cause of foot-drop.
* History of dementia, severely impaired cognition, communication or comprehension deficits.
* Presence of severe or frequent headaches
* History of Botulinum toxin (Botox) injection to either of the lower extremities within the 3 month period preceding study entry.
* Have other medical conditions or are taking medications that compromise ambulation or balance.
* Failure to meet established screening criteria for TMS or tDCS (i.e., TASS)
* Principal Investigator's or Medical Monitor's discretion not to include a participant.

Additional Exclusion Criteria for MRI Scan

* Claustrophobia, or the inability to lie still in a confined space
* Major medical disorders (e.g., HIV, cancer)
* Medications which may affect image quality (e.g., water pills)
* Magnetic metallic implants (such as screws, pins, shrapnel remnants, aneurysm clips, artificial heart valves, inner ear (cochlear) implants, artificial joints, and vascular stents), as these may heat, pull, or twist in the strong magnetic field of the MRI scanner
* Non-removable dental implants, such as braces or permanent retainers, as these will distort the MRI images we collect (note: filings, crowns, and silver or gold teeth are OK)
* Permanent makeup or tattoos with metallic dyes
* A positive pregnancy test (for females), since the effect of strong magnetic fields on the developing fetus remains unknown and inconclusive. (We will conduct a pregnancy test for all female participants on the day of the MRI scan.)
* Psychotic disorders (e.g., schizophrenia)
* Any other condition that the investigator believes might put the participant at risk

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mennemeier, PhD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - University of Central Arkansas, Conway, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via study advertisements and referrals from physical therapy clinics
Groups:
- Transcranial Direct Current Stim: tDCS will be applied using a DeluxeSoterix constant current stimulator with 5 x 5 cm (25cm2) carbon rubber electrodes (Covidien 664 REFX 2x2) applied to the scalp with 10-20 conductive paste. The anodal electrode will be placed over the lower extremity representation of primary motor cortex of the lesioned hemisphere [established during TMS motor threshold testing (Baseline Testing) and the functional MRI assessment]. The cathodal electrode will be placed over the contralateral motor cortex. During anodal tDCS, participants will receive 20 min at 2mA over motor cortex (with 30 seconds of ramp-up and ramp-down).
Period: Baseline
Arm/Group | Transcranial Direct Current Stim | Sham tDCS
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0
Period: One Week
Arm/Group | Transcranial Direct Current Stim | Sham tDCS
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0
Period: One Month
Arm/Group | Transcranial Direct Current Stim | Sham tDCS
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stim | Sham tDCS | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.9) | 45 (26.9) | 58.0 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ankle dorsiflexion angle during the swing phase of gait [Mean (Standard Deviation); unit: degrees] — Normal dorisflexion in mid-swing is 0. More than -5 degrees of plantar flexion is foot drop.
  degrees | -9.28 (3.10) | -0.19 (4.39) | -6.25 (10.21)
Slope of recruitment curve [Mean (Standard Deviation); unit: slope of regression line] — The recruitment curve consists of MEPs plotted for increasing intensities of TMS. The slope reflects the rate at which MEP values increase.
  slope of regression line | 7.24 (0.71) | 5.19 (.87) | 6.42 (2.09)
Stroke Impact Scale Score [Mean (Standard Deviation); unit: units on a scale] — Sixteen item scale. Range of scores is 16 to 80. High score means higher functioning.
  units on a scale | 53.0 (1.97) | 68.67 (2.78) | 58.22 (9.55)

OUTCOME MEASURES:

1. Primary Outcome: Ankle Dorsiflexion Angle. Change From Baseline in Ankle Dorsiflexion Angle During the Swing Phase of Gait
Description: Over ground laboratory assessments of gait: 1) Gait velocity and spatiotemporal gait parameters will be measured with the GAITRite system (CIR Systems, Inc., Havertown, PA) 28-35. 2) Hip, ankle, and knee angles during gait will be measured using the Simi Aktisys gait analysis system (Simi Reality Motion Systems; Postfach, Unterschleissheim Germany). LED markers are placed on the participant's lower extremity. Ankle, knee, and hip angle data is obtained simultaneously to evaluate motor strategies for overcoming gait impairments. Both types of data will be collected simultaneously as participants walk 10 meters across the GAITRite walkway at a self-selected speed for 5 repetitions.
Time Frame: Study week 1, and study weeks 5(± 5 days) and 8 (± 10 days).
Measure: Mean (Standard Error); unit: degrees
Groups:
- Active tDCS: Week 5 - Baseline.; Active tDCS: Week 8 - Baseline: tDCS will be applied using a DeluxeSoterix constant current stimulator with 5 x 5 cm (25cm2) carbon rubber electrodes (Covidien 664 REFX 2x2) applied to the scalp with 10-20 conductive paste. The anodal electrode will be placed over the lower extremity representation of primary motor cortex of the lesioned hemisphere [established during TMS motor threshold testing (Baseline Testing) and the functional MRI assessment]. The cathodal electrode will be placed over the contralateral motor cortex. During anodal tDCS, participants will receive 20 min at 2mA over motor cortex (with 30 seconds of ramp-up and ramp-down).
- Sham tDCS; Week 5 - Baseline.; Sham tDCS: Week 8 - Baseline.: Sham stimulation will be performed by turning the stimulator off after the initial sensory experience (30 seconds).
Arm/Group | Active tDCS: Week 5 - Baseline. | Active tDCS: Week 8 - Baseline | Sham tDCS; Week 5 - Baseline. | Sham tDCS: Week 8 - Baseline.
Number analyzed (Participants) | 4 | 4 | 2 | 2
degrees | 3.85 (7.60) | .18 (7.60) | -4.15 (10.74) | -1.60 (10.74)
Statistical Analysis 1: Comparison: Active tDCS: Week 5 - Baseline. vs Active tDCS: Week 8 - Baseline vs Sham tDCS; Week 5 - Baseline. vs Sham tDCS: Week 8 - Baseline; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = 9.10, Standard Error of Mean 5.37

2. Secondary Outcome: Slope of Recruitment Curve. Change From Baseline in the Slope of the Recruitment Curve Based on Motor Evoked Potentials (MEPs).
Description: A Magstim 200 super rapid2 stimulator with a 110 mm double cone coil will deliver stimulation. First, the TMS motor threshold (MT) will be established and the best location for eliciting MEPs from the contralesional and ipsilesional TA muscle will be tracked on the subject's MRI scan in Brainsight. Recruitment curves will be obtained as follows: 1) delivering ten, single TMS pulses beginning at 70% of MT, 2) increasing TMS intensity by 10% and repeating the process up to 160% of the MT or until a plateau in the recruitment curve is reached, 3) offline data processing will be performed with the Matlab curve fitting toolbox and 4) the threshold, slope, and MEPmax, and the goodness of fit (R2) will be calculated. A change in the slope of the recruitment curve will indicate change in cortical excitability.
Time Frame: Study week 1, and study weeks 5(± 5 days) and 8 (± 10 days).
Measure: Mean (Standard Error); unit: Slope of a regression line
Arm/Group | Active tDCS: Week 5 - Baseline. | Active tDCS: Week 8 - Baseline | Sham tDCS; Week 5 - Baseline. | Sham tDCS: Week 8 - Baseline.
Number analyzed (Participants) | 4 | 4 | 2 | 2
Slope of a regression line | .98 (1.73) | .89 (1.73) | -1.32 (2.12) | -1.84 (2.12)
Statistical Analysis 1: Comparison: Active tDCS: Week 5 - Baseline. vs Active tDCS: Week 8 - Baseline vs Sham tDCS; Week 5 - Baseline. vs Sham tDCS: Week 8 - Baseline; Test type: Superiority; p = .05, ANOVA; Mean Difference (Final Values) = -2.05, Standard Deviation 1.12

3. Secondary Outcome: Change From Baseline in Stroke Impact Scale Scores
Description: The Stroke Impact Scale-16 (SIS-16, completed by study team) is a standardized instrument 36-38 that assesses 3 functional domains in stroke patients including ADL / IADL, mobility, and social and occupational engagement. It consists of 64 - 5 point likert scale questions with a total score range of 64(lowest) to 320 (highest).
Time Frame: Study week 1, and study weeks 5(± 5 days) and 8 (± 10 days).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active tDCS: Week 5 - Baseline. | Active tDCS: Week 8 - Baseline | Sham tDCS; Week 5 - Baseline. | Sham tDCS: Week 8 - Baseline.
Number analyzed (Participants) | 4 | 4 | 2 | 2
units on a scale | 1.75 (4.82) | 1.25 (4.82) | 6.82 (.77) | 00. (6.80)
Statistical Analysis 1: Comparison: Active tDCS: Week 5 - Baseline. vs Active tDCS: Week 8 - Baseline vs Sham tDCS; Week 5 - Baseline. vs Sham tDCS: Week 8 - Baseline; Test type: Superiority; p = .05, ANOVA; Mean Difference (Final Values) = 15.67, Standard Deviation 3.41

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over a 2 year period
Arm/Group | Transcranial Direct Current Stim | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/4 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transcranial Direct Current Stim (N=4) | Sham tDCS (N=2)
headache (General disorders) | 2 | 0
Rolled ankle (Musculoskeletal and connective tissue disorders) | 1 | 0
knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
CABG surgery (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT01807637/Prot_SAP_000.pdf